CLINICAL TRIAL: NCT00565201
Title: Evaluation of BOTOX® (Botulinum Toxin Type A) in Combination With Rehabilitation Therapy for the Treatment of Wrist and Hand Muscle Overactivity in Post-Stroke Patients
Brief Title: Evaluation of BOTOX® With Rehabilitation Therapy for the Treatment of Wrist and Hand Spasticity in Post-Stroke Patients
Acronym: Botox/Rehab
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Steven L. Wolf, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00002727
Record Dates: First submitted 2007-11-20; First posted 2007-11-29 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Stroke
Keywords: Stroke, Cerebrovascular accident, Spasticity, Arm, Hand
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox and Rehab (Experimental): Patients will receive BOTOX® (100 to 360 U) injected into the any of the following muscles: 30-100U in the Flex. Dig. Sublimes (3 sites), 30-100U in the flex. Carpi Rad. (3 sites), 30- 100 U flex Carpi Ulnaris (3 sites), 30-100 U in the flex Dig Superficiali ( 3 sites), 25U Prontator Teres (1 site), 25 U Brachioradialis (1 site).
  Physical Rehabilitation: One hour session divided into 3 categories of treatment - 1.) Pre-functional/modalities for a general guideline of treatment; 2.)Repetitive task practice and strengthening; 3.)Functional activities - ADL and IADLs.
  Interventions: Drug: Botox and rehab
- Placebo and Rehab (Placebo Comparator): Patients will placebo saline (100 to 360 U) injected into any of the following muscles: 30-100U in the Flex. Dig. Sublimes (3 sites), 30-100U in the flex. Carpi Rad. (3 sites), 30- 100 U flex Carpi Ulnaris (3 sites), 30-100 U in the flex Dig Superficiali ( 3 sites), 25U Prontator Teres (1 site), 25 U Brachioradialis (1 site) followed by Physical Rehabilitation: One hour session divided into 3 categories of treatment - 1.) Pre-functional/modalities for a general guideline of treatment; 2.)Repetitive task practice and strengthening; 3.)Functional activities - ADL and IADLs.
  Interventions: Drug: Placebo and rehab

INTERVENTIONS:
Drug: Botox and rehab — Patients will BOTOX® (100 to 360 U) injected into any of the following muscles: 30-100U in the Flex. Dig. Sublimes (3 sites), 30-100U in the flex. Carpi Rad. (3 sites), 30- 100 U flex Carpi Ulnaris (3 sites), 30-100 U in the flex Dig Superficiali ( 3 sites), 25U Prontator Teres (1 site), 25 U Brachioradialis (1 site) followed by Physical Rehabilitation: One hour session divided into 3 categories of treatment - 1.) Pre-functional/modalities for a general guideline of treatment; 2.)Repetitive task practice and strengthening; 3.)Functional activities - ADL and IADLs.
  Arms: Botox and Rehab
Drug: Placebo and rehab — Patients will receive placebo saline (100 to 360 U) injected into any of the following muscles: 30-100U in the Flex. Dig. Sublimes (3 sites), 30-100U in the flex. Carpi Rad. (3 sites), 30- 100 U flex Carpi Ulnaris (3 sites), 30-100 U in the flex Dig Superficiali ( 3 sites), 25U Prontator Teres (1 site), 25 U Brachioradialis (1 site) followed by Physical Rehabilitation: One hour session divided into 3 categories of treatment - 1.) Pre-functional/modalities for a general guideline of treatment; 2.)Repetitive task practice and strengthening; 3.)Functional activities - ADL and IADLs.
  Arms: Placebo and Rehab

SUMMARY:
The present study is designed to determine the safety and effectiveness of injections of BOTOX® in spastic muscles of the arm and hand compared with injections of saline (which would do nothing) when combined with rehabilitation therapy for the improvement of active function tasks in post-stroke patients. Injections will be targeted to reduce common spasticity patterns of the arm and hand which include: bent elbow, palm down forearm, bent wrist, thumb-in-palm, clenched fist, and other hand deformities. This will be done only at Emory University. Neither the doctor injecting the drug nor the subject receiving the drug will know if they are getting BOTOX® or saline. Which type of injection the subject receives will be completely randomized (like flipping a coin). All subjects will have rehabilitation therapy after their injections. Subjects will be assessed at a total of 5 scheduled visits (qualification (Week 1), Injection (Week 2), Evaluations on Weeks 8, 10, and 14. All subjects will receive rehabilitation therapy immediately after their injections for 1 hour a day, 3-5 times a week, for 4 weeks. The results from this project will provide valuable data on the ability of BOTOX® and physical rehabilitation to provide effective treatment to spastic muscles of the arm and hand after stroke. This project has the potential to increase the availability of effective rehabilitation techniques to patients with stroke.

DETAILED DESCRIPTION:
After a stroke, patients commonly experience tightness in their affected arm from wrist and hand muscle overactivity called spasticity. Spasticity is difficult to manage with only one type of treatment. Usual treatments of spasticity are not very effective and may produce unwanted side effects. Untreated spasticity may result in muscular problems and decrease a patient's general ability to function and thus affect his/her quality of life.

BOTOX®, a botulinum toxin type A produced from Clostridium botulinum, blocks certain chemicals that cause spasticity. With appropriate injections of BOTOX® in the correct muscle, it can change the tightness in the muscle temporarily. Published reports indicate that several hundred adult patients with arm and/or leg spasticity of various causes (e.g., poststroke, multiple sclerosis and traumatic brain injury) have benefited from injections of BOTOX® in the spastic muscle. The efficacy of BOTOX® in patients with post-stroke spasticity in their arms and hands has been demonstrated in seven phase 2 placebo-controlled studies and two phase 3 studies.

The present study is designed to determine the safety and effectiveness of injections of BOTOX® in spastic muscles of the arm and hand compared with injections of saline (which would do nothing) when combined with rehabilitation therapy for the improvement of active function tasks in post-stroke patients. Injections will be targeted to reduce common spasticity patterns of the arm and hand which include: bent elbow, palm down forearm, bent wrist, thumb-in-palm, clenched fist, and other hand deformities. This will be done only at Emory University. Neither the doctor injecting the drug nor the subject receiving the drug will know if they are getting BOTOX® or saline. Which type of injection the subject receives will be completely randomized (like flipping a coin). All subjects will have rehabilitation therapy after their injections. Subjects will be assessed at a total of 5 scheduled visits (qualification (Week 1), Injection (Week 2), Evaluations on Weeks 8, 10, and 14. All subjects will receive rehabilitation therapy immediately after their injections for 1 hour a day, 3-5 times a week, for 4 weeks. The results from this project will provide valuable data on the ability of BOTOX® and physical rehabilitation to provide effective treatment to spastic muscles of the arm and hand after stroke. This project has the potential to increase the availability of effective rehabilitation techniques to patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years of age
* Written informed consent
* Written Authorization for Use and Release of Health and Research Study Information has been obtained
* Medically stable condition in the investigator's opinion
* History of stroke (hemorrhagic or ischemic) that resulted in a unilateral, upper-limb focal spasticity pattern of the wrist and fingers
* EMG evidence of volitionary activiation of wrist and finger extensor and flexor muscles
* Active range of motion (to be repeated 3 times by the patient): The ability to initiate wrist extension of at least 10 degrees from a fully flexed position with the forearm supported and stabilized in a pronated position. Active shoulder flexion and abduction to 45 degrees and no less than -30 degrees of elbow extension.
* Mini-Mental State Exam (MMSE) >24
* If on an anti-spasticity medication regiment at the time of qualification, the dose regimen must have been stable 1 month prior to study enrollment
* Ability to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* Time since neurological event resulting in upper limb spasticity less than 3 months or greater than 24 months
* Previous therapy with BOTOX® or any other botulinum toxin serotype for any condition within the last 12 months
* Phenol or alcohol block in the study limb within 6 months of study enrollment visit
* History (within 3 months of qualification) of or planned (during study period) casting of the study limb
* Current treatment with an intrathecal baclofen pump
* In the opinion of the investigator, profound atrophy of the muscles in the study limb that are targeted for injection
* Previous surgical intervention in the study limb, except for routine orthopedic repair for bone fractures, in the last 6 months
* Presence of fixed contracture of the study limb impairing functional activity
* Clinically significant inflammation or condition in the study limb that, in the investigator's opinion, could limit joint movement (other than stroke or spasticity)
* Clinically significant spasticity or contracture of the elbow (defined as an Ashworth score >3) or shoulder in the study limb, in the investigator's opinion would limit sue of the wrist and fingers
* Changes in oral spasticity medications within 30 days of enrollment (dose of anti-spasticity medications should remain the same during the study)
* Anticipated use of oral coagulants during the study
* Known allergy or sensitivity to the study medication or its components
* Infection or dermatological condition at anticipated injection sites
* Current participation in another clinical study or within 1 month of the enrollment visit
* Females who are pregnant, nursing, or planning a pregnancy during the study, or females of childbearing potential, not using a reliable means of contraception
* Anticipated use during the study of concurrent therapies for treatment of upper motor neuron syndrome (eg, acupuncture)
* Any medical condition that may put the patient at increased risk with exposure to BOTOX including diagnosed myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function
* Patient has a condition or is in a situation which in investigator's opinion may put the patient significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy
Arm Motor Ability Test | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy

SECONDARY OUTCOMES:
Stroke Impact Scale | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy
Modified Ashworth Scale | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy
Upper Extremity range of motion measurements | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy
Caregiver questionnaire | Baseline, Pre-therapy, Post-therapy, and 1 month after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Wolf, PhD, PT, Principal Investigator — Emory University; Byron Milton, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States